CLINICAL TRIAL: NCT05514665
Title: A Prospective Feasibility Study to Derive Novel Imaging Biomarker of Perinatal Brain Injury Based on Bedside Diffuse Optical Tomography in Neonates
Brief Title: Functional Imaging of Baby Brains
Acronym: FIBB
Status: Recruiting | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: NIF-22535
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-03

CONDITIONS: Hypoxia Ischemia, Cerebral; Hypoxia-Ischemia, Brain; Hypoxia Neonatal; Hypoxic-Ischemic Encephalopathy
Keywords: diffuse optical tomography; functional near-infrared spectroscopy; neuroimaging; functional connectivity; resting state networks
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neonates with perinatal hypoxic-ischemic brain injury: Neonates who are admitted to the Level III Neonatal Intensive Care Unit with a diagnosis of hypoxic ischemic encephalopathy will undergo diffuse optical tomography measurements prior to discharge from Neonatal Intensive Care Unit . Their developmental assessment will be performed at 6 months and 12 months postmenstrual age.
  Interventions: Device: Diffuse Optical Tomography

INTERVENTIONS:
Device: Diffuse Optical Tomography — Neonates once hemodynamically stable will undergo diffuse optical tomography measurements of functional brain connectivity at the bedside within 3-7 days after birth.

SUMMARY:
Infants are at risk of developing motor and cognitive neurodevelopmental disabilities as a sequelae to hypoxic-ischemic brain injury during the perinatal period. It is an ongoing challenge to predict the severity and extent of future developmental impairment during the neonatal period. This study will help test the feasibility of conducting a large-scale study that evaluates the role of diffuse optical tomography as a bedside neuroimaging tool in complementing the prognostic value of conventional and diffusion weighted MRI for predicting neurodevelopmental outcome in neonates with perinatal hypoxic-ischemic brain injury.

DETAILED DESCRIPTION:
Perinatal hypoxic-ischemic brain injury is a major cause of childhood disabilities including cerebral palsy, developmental delay, attention deficits, behavioral concerns, and learning disabilities. Accurate prediction of neurologic deficits in the neonatal period is difficult, especially the ability to predict later cognitive impairment and socio-emotional challenges. Many of these disabilities are manifested at school age when the child is beyond the critical time window of early brain development. Prognostic tools that help to identify neonates most at risk of developing neuro-deficits after perinatal asphyxia are needed and would enable targeted early intervention in infancy, when the developing brain is most amenable to positive changes and improve neurologic outcome. Currently, structural changes observed in MRI brain images are used to predict outcome. However, this modality does not provide information on brain function, nor is it a good prognostic marker of future neurocognitive outcome. Functional MRI (fMRI) is time-consuming and not commonly a part of clinical assessment of the neonates. Diffuse Optical Tomography (DOT) using near-infrared light has been applied in research settings to map the functional connections between key brain regions. This technology, although reported to be safe and reliable in small studies, has not been widely used in the neonatal clinical setting. This approach is based on the synchronous, spontaneous fluctuations of cerebral blood flow in different regions of the brain that are functionally, yet not necessarily anatomically connected. DOT combines the portability and cap-based scanning of EEG with spatial resolution high enough to create detailed cortical maps of the neonatal brain. Compared to MRI and fMRI brain imaging, DOT is portable, light weight, has high body motion tolerance, does not produce noise and does not require infant sedation. It has the potential to be a powerful bedside non-invasive clinical neuroimaging tool. Currently, the predictive accuracy of DOT based neonatal brain connectivity measures in prognosticating early childhood is unknown. This study aims to assess the feasibility of the processes that are key to the success of a large-scale prospective study aimed at investigating the prognostic value of bedside DOT derived biomarker in neonatal brain after perinatal hypoxic-ischemic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to the McMaster Children's Hospital Neonatal Intensive Care Unit with the diagnosis of hypoxic-ischemic encephalopathy will be considered for this study
* Gestational age of 35 weeks or greater
* Birth weight more than 1.8 Kg

Exclusion Criteria:

(i) suspected or confirmed congenital malformations, (ii) chromosomal anomalies, (iii) inborn errors of metabolism, (iv) congenital infections, (v) neonatal encephalopathy other than HIE, (vi) baby requires respiratory support in the form of CPAP, Mechanical ventilation, high flow nasal cannula and (vii) scalp injury or non-intact skin surface in the scalp

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A cohort of neonates admitted with clinical history suggestive of perinatal hypoxic-ischemic encephalopathy will be enrolled to the study, irrespective of whether they are considered eligible or ineligible for therapeutic hypothermia. The intervention (DOT measurement) will be conducted after therapeutic hypothermia is completed and neonate is considered hemodynamically stable to tolerate the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Consent rate | 12 months
  An eligible patient (parents or substitute decision makers) consents to the study
Rate of completion of study intervention | 12 months
  An enrolled patient receives DOT measurements taken within 7 days of life
Rate of successful data acquisition | 12 months
  An enrolled patient completes resting state DOT data acquisition within 45 mins without sedation
Rate of developmental follow up | 12 months
  An enrolled patient is assessed for neurological outcome at the age of 6 months and 12 months

SECONDARY OUTCOMES:
Resting state connectivity measures | 12 months
  Strength of network connectivity in pre-identified brain regions i.e somatosensory cortex and auditory cortex
First time-point developmental assessment | 6 months post menstrual age
  Assessed by parent-filled questionnaire using Ages and Stages Questionnaire-3 rd edition. Total score in each domain (Cognitive, Gross motor, Fine motor, Problem solving, Personal social) ranges from 0-60. Higher score is better.
Second time-point developmental assessment | 12 months post menstrual age
  Assessed by parent-filled questionnaire using Ages and Stages Questionnaire-3 rd edition. Total score in each domain (Cognitive, Gross motor, Fine motor, Problem solving, Personal social) ranges from 0-60. Higher score is better

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doria V, Beckmann CF, Arichi T, Merchant N, Groppo M, Turkheimer FE, Counsell SJ, Murgasova M, Aljabar P, Nunes RG, Larkman DJ, Rees G, Edwards AD. Emergence of resting state networks in the preterm human brain. Proc Natl Acad Sci U S A. 2010 Nov 16;107(46):20015-20. doi: 10.1073/pnas.1007921107. Epub 2010 Nov 1. PMID 21041625
- [Background] Gao W, Alcauter S, Elton A, Hernandez-Castillo CR, Smith JK, Ramirez J, Lin W. Functional Network Development During the First Year: Relative Sequence and Socioeconomic Correlations. Cereb Cortex. 2015 Sep;25(9):2919-28. doi: 10.1093/cercor/bhu088. Epub 2014 May 8. PMID 24812084
- [Background] Fransson P, Skiold B, Horsch S, Nordell A, Blennow M, Lagercrantz H, Aden U. Resting-state networks in the infant brain. Proc Natl Acad Sci U S A. 2007 Sep 25;104(39):15531-6. doi: 10.1073/pnas.0704380104. Epub 2007 Sep 18. PMID 17878310
- [Background] Gollenberg AL, Lynch CD, Jackson LW, McGuinness BM, Msall ME. Concurrent validity of the parent-completed Ages and Stages Questionnaires, 2nd Ed. with the Bayley Scales of Infant Development II in a low-risk sample. Child Care Health Dev. 2010 Jul;36(4):485-90. doi: 10.1111/j.1365-2214.2009.01041.x. Epub 2009 Dec 16. PMID 20030657
- [Background] Ferradal SL, Liao SM, Eggebrecht AT, Shimony JS, Inder TE, Culver JP, Smyser CD. Functional Imaging of the Developing Brain at the Bedside Using Diffuse Optical Tomography. Cereb Cortex. 2016 Apr;26(4):1558-68. doi: 10.1093/cercor/bhu320. Epub 2015 Jan 16. PMID 25595183
- [Background] Liao SM, Gregg NM, White BR, Zeff BW, Bjerkaas KA, Inder TE, Culver JP. Neonatal hemodynamic response to visual cortex activity: high-density near-infrared spectroscopy study. J Biomed Opt. 2010 Mar-Apr;15(2):026010. doi: 10.1117/1.3369809. PMID 20459255
- [Background] Niu H, Li Z, Liao X, Wang J, Zhao T, Shu N, Zhao X, He Y. Test-retest reliability of graph metrics in functional brain networks: a resting-state fNIRS study. PLoS One. 2013 Sep 9;8(9):e72425. doi: 10.1371/journal.pone.0072425. eCollection 2013. PMID 24039763
- [Background] Lee CW, Cooper RJ, Austin T. Diffuse optical tomography to investigate the newborn brain. Pediatr Res. 2017 Sep;82(3):376-386. doi: 10.1038/pr.2017.107. Epub 2017 May 31. PMID 28419082
- [Background] Smyser CD, Wheelock MD, Limbrick DD Jr, Neil JJ. Neonatal brain injury and aberrant connectivity. Neuroimage. 2019 Jan 15;185:609-623. doi: 10.1016/j.neuroimage.2018.07.057. Epub 2018 Jul 27. PMID 30059733
- [Background] Zhang X, Toronov V, Webb A. Simultaneous integrated diffuse optical tomography and functional magnetic resonance imaging of the human brain. Opt Express. 2005 Jul 11;13(14):5513-21. doi: 10.1364/opex.13.005513. PMID 19498547